CLINICAL TRIAL: NCT04177550
Title: Early Results of Empyema Thoracis Treatment in Children by Video-assisted Thoracoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nhan Pham Nguyen Hien (Other)
Collaborators: Ho Trung Cuong (Unknown); Trinh Nguyen Ha Vi (Unknown); Tran Nhu Quynh (Unknown); Vu Minh Thuy (Unknown); Nguyen Thi Tuong Lam (Unknown)
Responsible Party: Sponsor-Investigator, Nhan Pham Nguyen Hien, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: NT 62 72 07 35
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Empyema Thoracis in Children
Keywords: empyema thoracis; Thoracoscopic; VATS; Video-assisted Thoracoscopic Surgery; Pediatric Empyema Thoracis
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of study is to assess early results of Empyema Thoracis treatment in Children by Video-assisted Thoracoscopic Surgery

ELIGIBILITY:
Inclusion Criteria:

* All patients had empyema.
* All patients had been treated by Video-assisted Thoracoscopic Surgery in Children hospital 1 from 01/01/2015 to 30/04/2019.

Exclusion Criteria:

* The patient had empyema caused by Tuberculosis.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patient had empyema who treated by Video-assisted Thoracoscopic Surgery in Children hospital 1 from 01/01/2015 to 30/04/2019
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2019-12-21 (Estimated); Primary Completion 2019-12-21 (Estimated); Study Completion 2020-05-21 (Estimated)

PRIMARY OUTCOMES:
Recover | 2 hours
  Time of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Children hospital no.1, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
We will decide when the research is complete